CLINICAL TRIAL: NCT03652025
Title: The Effectiveness of Trans-catheter Foam Sclerotherapy of Pelvic and Atypical Lower Limb Varicosities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ahmadnaserhussein, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU777
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Intervention Model Description: premenopausal women with dull aching pain with ovarian point tenderness and post coital pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): perimenopausal women
  Interventions: Procedure: embolotherapy of incompetent gonadal and iliac veins

INTERVENTIONS:
Procedure: embolotherapy of incompetent gonadal and iliac veins — minimally invasive

SUMMARY:
pelvic congestion is the most recognized consequence of pelvi-perineal venous insufficiency .

chronic pelvic pain prevalence is about 26.6 %in egypt. this research is going to evaluate the effectiveness of foam sclerotherapy and to conclude diagnostic and therapeutic algorithm for this problem.

DETAILED DESCRIPTION:
this study includes clinical and imaging and interventional aspects. detailed history and comprehensive examination of the patient. duplex ultrasonography to detect pelvic varices and presence of reflux. renal and left iliac venogram is usually the first step in the evaluation of compressive syndrome. then cannulate the gonadal and internal iliac veins selectively. contrast medium injected , the incompetent gonadal veins are generally dilated and the contrast pools in the pelvis after injection. embolization by injecting afoam sclerosant as distally as possible to occlude the pelvic venous plexus using occlusion balloon proximal.

follow up assessment by VAS score and duplex imaging.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal women ovarian point tenderness post coital pain atypical lower limb varices

Exclusion Criteria:

* endometriosis diverticulitis fasciitis psychosexual dysfunction

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
The difference in pain score before and after therapy | one year
  validated analogue scoring of pain From 0 to 10 according to symptoms improvement